CLINICAL TRIAL: NCT05402098
Title: Comparative Evaluation of Outcome Following Endodontic Treatment Using Traditional Versus Conservative Access in Mandibular Molars With Symptomatic Irreversible Pulpitis: a Randomized Controlled Trial
Brief Title: Outcome Following Endodontic Treatment Using Traditional Access Versus Conservative Access
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A Ramani
Record Dates: First submitted 2022-05-29; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Pulpitis - Irreversible
Keywords: Irreversible pulpitis; Endodontic treatment; Traditional access; Conservative access; Contracted endodontic cavities

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endodontic treatment using traditional access (Active Comparator): Straight line access will be achieved following complete removal of pulp chamber roof
  Interventions: Procedure: Endodontic treatment using traditional access
- Endodontic treatment using conservative access (Experimental): Part of pulp chamber roof will be preserved and no efforts will be directed to achieve straight line access
  Interventions: Procedure: Endodontic treatment using conservative access

INTERVENTIONS:
Procedure: Endodontic treatment using traditional access — Endodontic treatment will be carried out following complete removal of pulp chamber roof and achieving straight line access
  Arms: Endodontic treatment using traditional access
Procedure: Endodontic treatment using conservative access — Endodontic treatment will be carried out following partial removal of pulp chamber roof, extended only to the extent which helps to locate all the orifices with no efforts will be made to achieve straight line access
  Arms: Endodontic treatment using conservative access

SUMMARY:
This study will compare the outcome of endodontic treatment using conservative or traditional access design in permanent molars with clinical signs indicative of irreversible pulpitis

DETAILED DESCRIPTION:
After thorough history and clinical and radio graphic examination, and confirmation of eligibility for the study, written informed consent will be obtained after explaining the procedure and its associated risks and benefits.

Clinical diagnosis of symptomatic irreversible pulpitis will be established based on a history of spontaneous pain or pain exacerbated by cold stimuli and lasting for a few seconds to several hours (lingering pain) compared to control teeth and which is reproducible using cold testing.

Once included, study subjects will be randomly allocated to either traditional access or conservative access group. Subsequently biomechanical preparation will be carried out using standard protocol with the use of rotary NiTi file system followed by root canal filling using gutta percha and zinc oxide eugenol sealer. Teeth will be restored using composite resin in the same appointment.

Pain analysis will be carried out preoperatively and postoperatively at every 24 hours till 7 days after intervention. All the subjects will be followed up for evaluation of success at 6 and 12 months from baseline.

ELIGIBILITY:
Inclusion Criteria:

* The patient should be ≥18 years of age.
* Restorable mandibular molars with extremely deep caries involving occlusal surface only
* Clinical diagnosis of symptomatic irreversible pulpitis with PAI score ≤2.
* Tooth should give positive response to pulp sensibility testing.
* Tooth with probing pocket depth and mobility are within normal limits.
* Non-contributory medical history.

Exclusion Criteria:

* Teeth with immature roots.
* No pulp exposure even after caries excavation.
* Teeth with signs of pulpal necrosis including sinus tract or swelling.
* Teeth with percussion sensitivity
* Positive history of antibiotic use in the past 1 month or requiring antibiotic prophylaxis
* Had taken analgesic in past 3 days
* Teeth with pathologic changes such as internal or external resorption
* Teeth with morphological variation
* Teeth with root canal calcification
* Teeth with fixed full coverage prosthesis

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Estimated)
Dates: Start 2022-05-12 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Clinical and radiographic success | Baseline to 12 Months
  CLINICAL SUCCESS CRITERIA:
  Absence of spontaneous pain, discomfort, swelling, sinus tract or tenderness to palpation or percussion.
  RADIOGRAPHIC SUCCESS CRITERIA:
  No pathosis evident on the radiograph such as root resorption, furcal pathosis or new periapical pathosis.
  Periapical Index score 1 or 2 according to Orstavic et al. Evaluation of both clinical and radiographic outcome is must for analyzing the actual success of therapeutic technique.
  Number of participants fulfilling both clinical as well as radiographic success criteria will be considered in success category.

SECONDARY OUTCOMES:
Pain analysis | Baseline to 7 days
  To assess incidence and intensity of pain postoperatively at every 24 hours till 7 days using Visual analogue Scale of 0 to 100 Millimeter line. Score 0 means no pain and Score 100 means maximum pain.

CONTACTS AND LOCATIONS:
Overall Officials: DR. ANKITA RAMANI, MDS, Principal Investigator — PGIDS, ROHTAK, HARYANA, INDIA-124001
Locations (1):
- Dr. Ankita Ramani, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No